CLINICAL TRIAL: NCT05608356
Title: Effect of Injectable Platelet-rich Fibrin (i-PRF) on the Rate of Orthodontic En Masse Retraction of Maxillary Anterior Teeth: A Randomized Controlled Clinical Trial
Brief Title: Effect of Injectable Platelet-rich Fibrin on the En Masse Retraction of Maxillary Anterior Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed magdy Mohamed Sabrah, PhD Candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: i-prf-en-masse-cu-2022-11-1
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Platelet-rich Fibrin
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: interventional group will receive injectable platelet rich fibrin intraligamentally distal to the right and left canines, and palatal to the upper 4 incisors, in three time points with 21 days interval, control group will receive sham injection instead.
Who Masked: Participant, Outcomes Assessor
Masking Description: Data assessment will be blinded as an assessor not participating in the study will be responsible for measuring the rate of en masse retraction, as the patient name could be hidden during data analysis. The models will be coded with numbers assigned to the participants, and will be sent to an assessor not participating in the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Intervention group subjects will receive injectable platelet rich fibrin (i-prf) . The (i-prf) will be injected in the periodontal ligament of maxillary anterior teeth during en masse retraction.The injection sites will be the sites of bone compression to target the surfaces of the bone where osteoclastogenesis and bone resorption occurs during en masse retraction.
  Considering that the obtained (i-prf) after centrifuging would be 4 ml, 1 ml will be injected intraligamentally distal to the right and left canines, and 0.5 ml will be injected intraligamentally palatal to each incisor. The study group will receive i-PRF intraligamentally in the periodontal ligament space of the maxillary six anterior teeth three times as follow, just before anterior teeth retraction, and after 21 days of the retraction, and after 42 days of the retraction. Before each time of injection, an anesthetic solution will be administered for pain control.
  Interventions: Biological: injectable platelet rich fibrin(i-prf)
- control group (Sham Comparator): Subjects in the control group will only receive sham (placebo) injection three successive times with and interval of 21days between each injection, similar to the timepoints of (i-prf) injection in the intervention group. Also the sites of injection will be similar to the sites of injection of the intervention group; 1 ml of the placebo agent will be injected intraligamentally distal to the right and left canines, and 0.5 ml will be injected intraligamentally palatal to each incisor. An anesthetic solution will be administered for pain control before the administration of the sham injections.
  Interventions: Drug: Sham Injection

INTERVENTIONS:
Biological: injectable platelet rich fibrin(i-prf) — I-prf is a second-generation PRP where autologous platelets and leukocytes are present in a complex fibrin matrix and can be obtained from blood using low-speed centrifugation without adding anticoagulants.
  Arms: intervention group
Drug: Sham Injection — Sham injection as a placebo injection
  Arms: control group

SUMMARY:
The aim of this study is to investigate the effect of local injection of injectable platelet rich fibrin (i-PRF) on the rate of orthodontic en masse retraction of anterior teeth clinically and to report any associated pain as well.

DETAILED DESCRIPTION:
Trial will be carried on 2 groups, each involve 13 participants with a total of 26 participants.

1. Subject examination to ensure he/she meets the eligibility criteria of the research.
2. Leveling and alignment using fixed orthodontic appliance.
3. Upper first premolars extraction as a part of the orthodontic treatment planning.
4. With the starting of en masse retraction, injection of the (i-prf) obtained from venous sample palatally and distally to the anterior teeth in the intervention group, and sham injection in the control group. The injection in both groups will be done just before retraction, 21 and 42 days after beginning of retraction Rate of en masse retraction will be calculated for patients in both groups at the monthly basis for for months after starting en masse retraction, data will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

1. Orthodontic patients with and age range (16 - 30) years.
2. Protruded upper anterior teeth requiring extraction of first premolars and anterior teeth retraction; Angle class I mal-occlusion with bi-alveolar dental protrusions or class II division 1.
3. Patients with full permanent dentition (with the exception of third molars).
4. Healthy dental and periodontal condition with good oral hygiene

Exclusion Criteria:

1. Patients with extensive restorations on the anterior teeth.
2. Subjects taking medication affecting inflammatory process of the orthodontic tissue reaction.
3. History of previous orthodontic treatment or trauma to the anterior teeth.
4. Syndromic patients and patients with systemic diseases.
5. Poor oral hygiene or periodontal diseases.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of En masse retraction | 4 months
  Alginate impression will be taken for each participant to obtain a plaster model obtained at five time points: before incisor retraction (T0), after one month (T1), after two months (T2), after three months(T3), and after four months (T4) of retraction. The models will be coded with numbers assigned to the participants, and will be sent to an assessor not participating in the research. In both groups, the amount of space closure will be calculated by a digital caliper in millimeters for each time point (T) and averaged for right and left sides.

SECONDARY OUTCOMES:
Associated Pain | 4 months
  Pain will be assessed using a visual analogue scale questionnaire that will be completed by the patient starting from the day following i-prf injection in the intervention group or the sham injection in the control group, the questionnaire will be repeated every month until the fourth month

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No